CLINICAL TRIAL: NCT04821986
Title: Oral Manifestation in Patients With SARS-CoV2 Infection.
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Other Study IDs: Oral SARS-CoV2
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV Infection
Keywords: oral Manifestation; SARS-CoV2; prevelance
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Oral Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The oral cavity is particularly susceptible to viral infection with several viruses such as herpes simplex virus, cytomegalovirus and Zika virus because of its structures, especially salivary glands and soft tissues Moreover, oral mucosa can be affected by secondary pathological process of a bacterial or fungal nature due to viral immunosuppression. The oral cavity could be considered a "biological barometer" of both viral infection and viral immunosuppression advancement .

DETAILED DESCRIPTION:
The SARS-Cov2 virus was identified in china at the end of 2019 and spread worldwide causing a global pandemic. Current research showed that SARS-Cov2 virus invades human cells via the receptor angiotensin-converting enzyme 2 (ACE2) through scRNA-seq data analyses. The study identified the organs that are at risk and are vulnerable to SARS-CoV-2 infection. Therefore, cells with ACE2 receptor distribution may become host cells for the virus and cause inflammatory response in related organs and tissues, such as the tongue mucosa and salivary glands. These results suggest that oral mucosa could be a target of SARS-CoV-2 infection .

Although many authors reported the presence of oral lesion associated with SARS-CoV2 infection, the prevalence of the oral manifestation and the range of oral manifestation are still unknown. Further studies are necessary to better understanding of the symptoms of the SARS-CoV2 virus in order to faster detection. A multidisciplinary team following the patients could be the key in treatment of the infection and faster recovery.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of SARS-CoV2 with PCR.
* Age range from 18-60 years old

Exclusion Criteria:

* Pregnancy or contraceptive pills
* Lactation
* Any auto-immune disease that could affect the oral mucosa
* On any neoplastic therapy.
* Uncontrolled diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with SARS-CoV2 infection confirmed with PCR will be recruited form 3 different isolation hospitals at Ministry of health and population. Patient selection will be based on certain inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
oral manifestation | one week
  describe the patient oral manifestation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] La Rosa GRM, Libra M, De Pasquale R, Ferlito S, Pedulla E. Association of Viral Infections With Oral Cavity Lesions: Role of SARS-CoV-2 Infection. Front Med (Lausanne). 2021 Jan 14;7:571214. doi: 10.3389/fmed.2020.571214. eCollection 2020. PMID 33521007
- [Result] Halboub E, Al-Maweri SA, Alanazi RH, Qaid NM, Abdulrab S. Orofacial manifestations of COVID-19: a brief review of the published literature. Braz Oral Res. 2020 Oct 30;34:e124. doi: 10.1590/1807-3107bor-2020.vol34.0124. eCollection 2020. PMID 33146320